CLINICAL TRIAL: NCT02190487
Title: Incidence and Risk Factors of Acute Kidney Injury After Thoracic Aortic Surgery Due to Dissection
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2011-0076
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Dissection of Thoracic Aorta
MeSH Terms: conditions — Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAS group: patients who had thoracic aortic surgery due to dissection

SUMMARY:
Acute kidney injury (AKI) is one of the most frequently encountered and prognostically significant complications after cardiovascular surgery. However, there is no definitive treatment to intervene after development of AKI, therefore, preventive strategy has been the major issue. By this time, incidence of AKI after cardiovascular surgery has been reported 3-50% based on the studies with various definition of AKI and different patient cohorts. Development of unified definition for AKI in the early 2000s opened a new era in AKI study.

According to the previous studies, aortic surgery, especially thoracic aortic surgery was known to be highly prevalent of AKI, which was considered to be caused by use of total circulatory arrest (TCA), relatively high number of emergency cases, combined malperfusion syndrome before surgery and relatively complicated surgical procedure. However, there has not been many studies of AKI in thoracic aortic surgery because of its low incidence and urgent clinical presentation of aortic pathology, which hinder large randomized controlled study. Moreover, there are conflicting reports of incidence and risk factors of AKI after thoracic aortic surgery, no conclusive result has been made. Therefore, this study was designed to investigate the incidence and risk factors after thoracic aortic surgery only due to dissection.

ELIGIBILITY:
Inclusion Criteria:

* thoracic aortic surgery due to dissection

Exclusion Criteria:

* chronic kidney disease on renal replacement therapy before surgery
* death during or within 24 hours after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had thoracic aortic surgery due to dissection
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
incidence of acute kidney injury based of RIFLE criteria | upto 7 days after surgery
  serum creatinine, GFR were retrospectively retrieved from electrical medical record upto 7days after surgery.

SECONDARY OUTCOMES:
Risk factors of acute kidney injury | after diagnosis of acute kidney injury after operation (usually within 7 days after operation)
  * age, sex, comorbidities
  * serum creatinine, hemoglobin,mean arterial blood pressure
  * CPB duration, aorta cross clamping duration, total circulatory arrest duration, operative procedures performed, amount of transfused blood components
  * serum creatinine upto 7 days after surgery, mean arterial pressure, cardiac index, amount of transfused blood components in intensive care unit, ventiltor duration, ICU stay duration, renal replacement therapy, 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yon Hee Shim, Study Director — Yonsei University
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea